CLINICAL TRIAL: NCT05289622
Title: Single-arm Prospectus Study to Evaluate the Safety and Security of the Expandable Valve Stent, Approach Technique and Its Implantation in the Pulmonary Position
Brief Title: Stent Implantation of Polyurethane Expandable Valve, by Catheter, in Patients With Pulmonary Valve Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Miguel Angel Maluf (Other)
Collaborators: SYNTHETIC HEART TECHNOLOGY (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Miguel Angel Maluf, Principal Investigator, Hospital Alemão Oswaldo Cruz
Organization: Hospital Alemão Oswaldo Cruz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 43624621.7.0000.0070
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Valvulopathy
Keywords: pulmonary valve dysfunction; pulmonary valvulopathy; Stent implant; Pulmonary valve disorders; Polyurethane Expandable Valve Stent; Tetralogy of Fallot; Cardiac insufficiency; right ventricular dysfunction; Pulmonary Valve Insufficiency; heart diseases; Prosthesis
MeSH Terms: conditions — Heart Valve Diseases; Tetralogy of Fallot; Heart Failure; Ventricular Dysfunction, Right; Pulmonary Valve Insufficiency; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, Single Arm Safety and Efficacy Study to evaluate the expandable polyurethane valve in the pulmonary position, in 5 patients over 18 years of age, with pulmonary valve dysfunction and moderate to severe impairment of cardiac ventricular function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Polyurethane expandable valve stent implant surgery (Experimental): Valve stent implantation will be performed under general anesthesia with transesophageal echocardiography monitoring, with thoracotomy approach median and circulation aid extracorporeal.
  Interventions: Device: Polyurethane expandable valve stent implant

INTERVENTIONS:
Device: Polyurethane expandable valve stent implant — The baseline assessment of patients will include the admission of patients and the performance of preoperative exams (cardiological imaging for the correct selection). An estimated surgery time of 5 hours. During the entire procedure, patients will be under general anesthesia and controlled mechanical ventilation. The material collected in the laboratory will be processed, the result released and discarded. After the patient enters the operating room, hemodynamic monitoring, ECG, arterial saturation, with peripheral sensor, central venous access with double lumen catheter will be carried out; blood pressure monitoring by radial artery puncture, bladder catheter and thermometer in the nasopharynx and rectum. After preoperative preparation, patients will undergo a surgical approach by median thoracotomy and installation of the Cardiopulmonary bypass (ECC) circuit, by placing a cannula in the ascending aorta, Superior Vena Cava (SVC) and Inferior Vena Cava (IVC).

SUMMARY:
Prospective Study, Single Arm to evaluate the safety and efficacy of polyurethane expandable valve implantation in the pulmonary position, in 5 patients over 18 years of age, with pulmonary valve dysfunction and moderate to severe impairment of Right Ventricular function. During throughout the study, safety parameters related to valve operation will be evaluated (patient's Functional Class), in addition to the occurrence of Serious Adverse Events. After the procedure, the patient must be hospitalized in the Intensive Care Unit until the complete hemodynamic stabilization and normalization of lung function and in good general condition (2 to 3 days of stay) and then transferred to the ward (2 to 3 days and stay) before hospital discharge. A formal Statistical Analysis Plan (SAP) will be developed and finalized before closing the database. Full details of data presentations and analysis will be provided in SAP.

Additional statistical analyses, other than those described in this section, may be performed if deemed appropriate and included in SAP. Any deviations from the final analysis plan or what is presented in the protocol will be discussed in the final study report. No formal inferential statistics will be applied to the data collected in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Pulmonary valve dysfunction and moderate to severe impairment of Right Ventricle function;
* Functional Class II to IV New York Heart Association (NYHA) classification of heart failure.

Exclusion Criteria:

* Impairment of cardiovascular function;
* Neurological impairment;
* Syndromes without prognosis or survival of less than 1 year;
* Carriers of infection undergoing medical treatment;
* Patients undergoing artificial life support;
* Known hypersensitivity to aspirin or heparin;
* Positive urine or serum test for pregnancy in female patients of reproductive age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Regurgitation After Polyurethane Expandable Valve Stent Implant Surgery | 6 months
  if there are changes in pulmonary regurgitation (PR): discreet or less (≤2+) on transthoracic echocardiogram (TTE).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Maluf, Principal Investigator — Hospital Alemão Oswaldo Cruz
Locations (1):
- Hospital Alemão Oswaldo Cruz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
A representative appointed by the study sponsor, regulatory authorities, or other auditing bodies whose job it is to verify that the research is being conducted properly may review any study data and records maintained by the study physician at the research site only, maintaining the privacy and anonymity of each participant.